CLINICAL TRIAL: NCT02140528
Title: Evaluation the Safety and Efficacy of Allogeneic Mesenchymal Stem Cell Transplantation in Tibial Closed Diaphyseal Fractures
Brief Title: Allogeneic Mesenchymal Stem Cell Transplantation in Tibial Closed Diaphyseal Fractures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Royan-Bone-012
Record Dates: First submitted 2014-05-14; First posted 2014-05-16 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Tibial Fracture
Keywords: Allogenic adipose derived mesenchymal stem cell tibial fracture
MeSH Terms: conditions — Tibial Fractures | interventions — Stem Cell Transplantation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mesenchymal stem cell receipients (Experimental): Transplantation of allogenic adipose derived mesenchymal stem cells in patients with tibial fracture.
  Interventions: Biological: Mesenchymal stem cell injection
- Placebo (Placebo Comparator): Placebo injection in the site of fracture in patients with tibia fracture.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Mesenchymal stem cell injection — Injection of adipose derived mesenchymal stem cell in the site of tibia fracture .
  Other Names: stem cell transplantation
  Arms: Mesenchymal stem cell receipients
Biological: Placebo
  Arms: Placebo

SUMMARY:
This study is a case-control prospective, clinal trial to assess the safety and efficacy of the allogeneic adipose derived mesenchymal stem cell transplantation on the healing of recent tibial fracture in 40 patients.

DETAILED DESCRIPTION:
In this study all eligible patients divided in 2 group.20 patients received allogeneic adipose derived mesenchymal stem cell in the fractured site (case group) and other patients received the placebo in the fractured site (control group) .

To assess the outcomes, we will evaluate the patients at 2, 6 weeks and 3, 6 months after transplantation by: X-ray, BMD , VAS and biochemical analysis with laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years
* The presence of tibial fracture based on X ray
* tibial fracture is limited to diaphysial

Exclusion Criteria:

* Addiction
* Pregnancy
* liver or kidney disease or uncontrolled diabetes or heart and lung disease
* immune deficiency

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Number of patients with union after transplantation of mesenchymal stem cell in case group in comparison with control group | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Nasser Aghdami, MD,PhD, Study Director — Head of regenerative medicine department &cell therapy center of Royan Institute; Mohsen Emaddedin, MD, Study Director — Department or regenerative medicine of Royan Institute.; Aziz Ahmadi, MD, Principal Investigator — Scientific board of Iranian Orthopedic Association; Maedeh Ghorbani, MD, Principal Investigator — Department of Regenerative Medicine; Afshin Farhadi, MD, Principal Investigator — Scientific board of Iranian Orthopedic Association
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- See also: Related Info — http://Royaninstitute.org